CLINICAL TRIAL: NCT00290706
Title: A Phase I/II Trial of Combination Bortezomib (VELCADE) and Gemcitabine Therapy for Patients With Relapsed or Refractory Aggressive B- and T-cell Non-Hodgkin's Lymphoma
Brief Title: A Phase I/II Trial of VELCADE & Gemcitabine for Patients With Relapsed or Refractory Aggressive B- and T-cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed per Data Monitoring Committee due to lack of efficacy
Sponsor: Northwestern University (Other)
Collaborators: Eli Lilly and Company (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 04H4; NU 04H4 (Other: Northwestern University); VEL-03-082; STU00007425 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 3 follicular lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Bortezomib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine 800 mg/m2 + Bortezomib IVP over 3-5 seconds (Experimental): Gemcitabine dose of 800 mg/m2 over 30 minutes followed by Bortezomib IVP given over 3-5 seconds on day 1 and day 15 of each cycle every 28 days for up to 8 cycles.
  Interventions: Drug: bortezomib; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: bortezomib — Bortezomib 1.6mg/m2 on days 1 and 15 of each cycle, given over 3-5 seconds on day 1 and day 15 of each cycle every 28 days for up to 8 cycles.
  Other Names: Velcade®; PS-341
Drug: gemcitabine hydrochloride — Gemcitabine dose of 800 mg/m2 over 30 minutes on day 1 and day 15 of each cycle every 28 days for up to 8 cycles.
  Other Names: Gemzar®

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine together with bortezomib may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of bortezomib when given together with gemcitabine and to see how well they work in treating patients with relapsed or refractory B-cell or T-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate (complete and partial remission) in patients with relapsed or refractory aggressive B- or T-cell non-Hodgkin's lymphoma treated with gemcitabine hydrochloride and bortezomib.
* Determine the maximum tolerated dose of bortezomib when administered with gemcitabine hydrochloride in these patients.

Secondary

* Determine the time to treatment failure, duration of response, and overall survival of patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.

OUTLINE: This is a phase I, dose-escalation study of bortezomib followed by a phase II, open-label study.

* Phase I: Patients receive gemcitabine hydrochloride IV over 30 minutes and bortezomib IV over 3-5 seconds on days 1 and 8. Treatment repeats every 21 days for up to 9 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 6 patients experience dose-limiting toxicity (DLT) OR the dose that at which 2 of 6 patients experience DLT.

* Phase II: Patients receive gemcitabine hydrochloride and bortezomib as in phase I at the MTD.

After completion of study therapy, patients are followed periodically for 3 years.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B- or T-cell non-Hodgkin's lymphoma (NHL)

  * Intermediate histology B-cell NHL, including any of the following:

    * Diffuse large B-cell lymphoma
    * Transformed large cell lymphoma
  * Any T-cell NHL histology
  * Cutaneous T-cell lymphoma (CTCL) or mycosis fungoides (MF) allowed
* Relapsed or refractory disease, defined as disease progressed after prior complete remission (CR), partial remission (PR), or stable disease (SD) to last therapy OR failure to achieve CR, PR, or SD after completion of last therapy
* Must have received 1-3 prior therapeutic regimens

  * Cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone (CHOP) AND cyclophosphamide, vincristine, and prednisone (CVP) OR CHOP with rituximab (CHOP-R) AND CVP with rituximab (CVP-R) is considered 1 regimen
  * Monoclonal antibody (e.g., rituximab) given as maintenance therapy is considered 1 regimen
  * Salvage chemotherapy followed by an autologous stem cell transplant is considered 1 regimen
  * No more than 7 prior therapeutic regimens for patients with CTCL or MF
* No mantle cell lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

  * At least 50,000/mm^3 if documented bone marrow involvement
* Hemoglobin ≥ 8.0 g/dL
* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* Bilirubin ≤ 2 times ULN
* Creatinine ≤ 2.0 mg/dL
* No known history of HIV infection
* No other active infection
* No uncontrolled hypertension
* No peripheral neuropathy ≥ grade 2 within the past 2 weeks
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No acute ischemia or active conduction system abnormalities by ECG
* No hypersensitivity to bortezomib, boron, or mannitol
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier-method contraception
* No serious medical or psychiatric illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

* Prior autologous and/or allogeneic stem cell transplantation allowed
* More than 3 weeks since prior chemotherapy, radiotherapy, or immunotherapy
* More than 3 weeks since prior systemic biologic anticancer therapy
* More than 3 weeks since prior systemic corticosteroids (e.g., oral prednisone > 10 mg per day)
* More than 2 weeks since prior investigational drug
* No prior bortezomib or gemcitabine hydrochloride
* No other concurrent systemic cytotoxic chemotherapy or investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-04-07 (Actual); Primary Completion 2011-02-11 (Actual); Study Completion 2012-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Gordon, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual to phase I on September 26, 2005 with first patient treated April 7 2006.The study was closed on October 17 2007 to phase I and opened to phase II on December 18 2007. The study closed permanently March 9 2011 with a total accrual of 32 patients treated on the study before reaching the total accrual goal.
Groups:
- Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.3 mg/m2: Patients are treated with Gemcitabine 800mg/m2 IV over 30 minutes and Bortezomib 1.3 mg/m2 IVP over 3-5 seconds on Day 1 and Day 8 of a 28 day Cycle for up to 8 cycles of treatment.
- Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2; Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D8: Patients are treated with Gemcitabine 800mg/m2 IV over 30 minutes and Bortezomib 1.6 mg/m2 IVP over 3-5 seconds on Day 1 and Day 8 of a 28 day Cycle for up to 8 cycles of treatment.
- Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D15: Patients are treated with Gemcitabine 800mg/m2 IV over 30 minutes and Bortezomib 1.6 mg/m2 IVP over 3-5 seconds on Day 1 and Day 15 of a 28 day Cycle for up to 8 cycles of treatment.
Period: Overall Study
Arm/Group | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.3 mg/m2 | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D8 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D15
Started | 5 | 6 | 7 | 14
Attempted1st Cycle (DLT period in phase I (Cohort 1 and Cohort 2) =20 days post Cycle 1) | 5 | 6 | 7 | 14
Reached 1st Response/Cycle 3 | 0 | 0 | 1 | 2
Completed | 0 | 0 | 1 | 2
Not Completed | 5 | 6 | 6 | 12
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 5 | 4 | 10
Not completed — Adverse Event | 0 | 1 | 2 | 0
Not completed — Receive auto transplant or radiation | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.3 mg/m2 | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D8 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D15 | Total
Number analyzed (Participants) | 5 | 6 | 7 | 14 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 5 | 9 | 22
  >=65 years | 2 | 1 | 2 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 4 | 5 | 14
  Male | 4 | 2 | 3 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 5 | 6 | 6 | 12 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 1 | 5
  White | 5 | 4 | 5 | 11 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 7 | 14 | 32

OUTCOME MEASURES:

1. Primary Outcome: Response Rate in Patients With Relapsed or Refractory B- and T-cell NHL With Gemcitabine and Bortezomib Combination Treatment.
Description: Response rate in patients with relapsed or refractory B- and T-cell NHL with Gemcitabine and Bortezomib combination treatment will be defined as the number of patients with Complete Remission [CR] and Partial Remission [PR]. CT scans at screening and after completing cycle 3, cycle 6 and 30 days after Cycle 8 assessed by the Response Criteria for Non-hodgkins Lymphoma will be used to determine response where:
  CR=Complete disappearance of all detectable clinical and radiographic evidence of disease PR=> 50% decrease in SPD of the six largest dominant nodes or nodal masses
Time Frame: At screening and after completing cycle 3, cycle 6 and 30 days after Cycle 8
Population: Patients must complete 3 cycles of treatment to be evaluable for this outcome measure. Only 3 patients reached Cycle 3 and the study closed before accrual was met due to lack of efficacy. Below shows response of patients that reached Cycle 3 and is not a reflection of response rate.
Measure: Number; unit: participants
Arm/Group | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.3 mg/m2 | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D8 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D15
Number analyzed (Participants) | 0 | 0 | 1 | 2
participants |  |  | 1 | 2

2. Secondary Outcome: Time to Treatment Failure and Duration of Response
Description: Time to treatment failure and duration of response will be measured by CT Scan at screening and after completing cycle 3, cycle 6 and 30 days after cycle 8, then every 6 months for 3 years
Time Frame: At screening and after completing cycle 3, cycle 6 and 30 days after cycle 8, then every 6 months for 3 years
Population: Study was terminated due to lack of efficacy. Data not collected for analysis of outcome measure.
Arm/Group | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.3 mg/m2 | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D8 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D15
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival will be evaluated every 6 months while on treatment and then every 6 months while off of treatment for up to 3 years
Time Frame: Every 6 months while on treatment and then every 6 months while off of treatment for up to 3 years
Population: The study was terminated early due to lack of efficacy. Data not collect for analysis of this outcome measure.
Groups:
- Gemcitabine 800 mg/m2 + Bortezomib IVP Over 3-5 Seconds: Gemcitabine dose of 800 mg/m2 over 30 minutes followed by Bortezomib IVP given over 3-5 seconds on either Day 1/Day 8 or Day 1/Day 15 of each cycle every 28 days for up to 8 cycles.
  Bortezomib: Bortezomib either 1.3 mg/m2 or 1.6mg/m2 on either Day 1/Day 8 or Day 1/Day 15 of each cycle, given over 3-5 seconds every 28 days for up to 8 cycles.
  Gemcitabine hydrochloride: Gemcitabine dose of 800 mg/m2 over 30 minutes on either Day 1/Day 8 or Day 1/Day 15 of each cycle every 28 days for up to 8 cycles.
Arm/Group | Gemcitabine 800 mg/m2 + Bortezomib IVP Over 3-5 Seconds
Number analyzed (Participants) | 0

4. Secondary Outcome: Evaluate Safety and Tolerability of Bortezomib and Gemcitabine Therapy
Description: Safety and tolerability of the study drugs will be assessed on Day 1 and on either Day 8 or Day 15 of each treatment cycle (1 Cycle - 28 days) while on active treatment; and 30 days post last treatment. Adverse Events that are experienced by patients, determined to be either grade 3 or grade 4 and at least possibly related to at least one of the study drugs as assessed according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0) will be collected. In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: During treatment through a maximum of 8 Cycles (1 Cycle = 28 Days) and 30 days post last treatment
Population: The study was terminated before total accrual was met due to lack of efficacy. Data was not collected for analysis for this outcome measure
Arm/Group | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.3 mg/m2 | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D8 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D15
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment through 30 days post treatment. The study was designed for a maximum of 8 Cycles of treatment (1 Cycle = 28 days) and the range of cycles attemted by any patient was 1 - 8.
Arm/Group | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.3 mg/m2 | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D8 | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D15
All-Cause Mortality (participants affected / at risk) | 5/5 | 6/6 | 7/7 | 11/14
Serious Adverse Events (participants affected / at risk) | 4/5 | 2/6 | 3/7 | 6/14
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 7/7 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.3 mg/m2 (N=5) | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 (N=6) | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D8 (N=7) | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D15 (N=14)
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Multi organ failure - death (General disorders) | 1 | 0 | 0 | 0
Progressive disease - death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 2
Fever (General disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pneumonia leading to death (Infections and infestations) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypertension (Cardiac disorders) | 0 | 1 | 0 | 0
Infection NOS (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 — Patient also with pneumonia during this event
Bacteremia (Infections and infestations) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Rectal bleeding (Renal and urinary disorders) | 0 | 0 | 0 | 1
Neutropenia (Infections and infestations) | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 — Patients also with Thrombocytopenia during this event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.3 mg/m2 (N=5) | Cohort 1 -Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 (N=6) | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D8 (N=7) | Phase II Gemcitabine 800 mg/m2 + Bortezomib 1.6 mg/m2 D1+D15 (N=14)
Hemoglobin decreased (Anemia) (Blood and lymphatic system disorders) | 4 | 3 | 5 | 9
Neutrophil decreased (neutropenia) (Blood and lymphatic system disorders) | 2 | 2 | 3 | 1
Leukocytes (Total white blood cells) (Blood and lymphatic system disorders) | 3 | 3 | 3 | 4
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 3 | 2 | 4 | 3
Platelet Decrease (Thrombocytopenia) (Blood and lymphatic system disorders) | 4 | 3 | 5 | 5
Hypertension (Cardiac disorders) | 0 | 2 | 0 | 1
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 2
Fatigue (General disorders) | 4 | 4 | 3 | 8
Fever (General disorders) | 3 | 2 | 2 | 1
Sweating (General disorders) | 1 | 0 | 0 | 1
Weight Loss (General disorders) | 0 | 1 | 0 | 1
Weight gain (General disorders) | 0 | 0 | 0 | 2
Skin (Not otherwise specified) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nasal Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Shingles (Infections and infestations) | 0 | 0 | 0 | 1
Hot flashes/Flashes (Endocrine disorders) | 0 | 0 | 0 | 1
Anorexia (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Dehydration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 1 | 5
Abdominal distension/bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Heartburn) (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 7
Dysgeusia (Taste Alteration) (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 4
Hemorrhage - Urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bruising (General disorders) | 1 | 0 | 0 | 0
Angular Cheilitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Infection in Leg (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sinus Infection (Infections and infestations) | 0 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Oral Ulcer (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Not otherwise specified) (Infections and infestations) | 0 | 0 | 2 | 0
Edema (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0
Edema in Limbs (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
Edema in Head and Neck (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Increased LDH (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Alkaline Phosphatase (Metabolism and nutrition disorders) | 2 | 3 | 1 | 3
Transaminase Increased (Metabolism and nutrition disorders) | 1 | 3 | 1 | 3
ALT Increased (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
AST Increased (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Albumin, Serum-Low (Metabolism and nutrition disorders) | 2 | 2 | 1 | 3
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Bicarbonate-Low (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Creatinine (Metabolism and nutrition disorders) | 3 | 2 | 1 | 2
Calcium, Serum High (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Glucose, Serum-High (Metabolism and nutrition disorders) | 4 | 1 | 1 | 7
Glucose, Serum-Low (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Magnesium, Serum-Low (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3
Phosphate, Serum-Low (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Potassium, Serum-High (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Potassium, Serum-Low (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Sodium, Serum-High (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Sodium, Serum-Low (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Uric Acid, Serum-High (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Sensory Neuropathy (Nervous system disorders) | 1 | 1 | 1 | 8
Pain (Nervous system disorders) | 0 | 0 | 0 | 1
Confusion (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in Throat (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pain in Abdomen (Not otherwise specified) (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Pain in Back (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in Extremities (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pain in Bones (General disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 1
Pain (Not otherwise specified) (General disorders) | 0 | 2 | 1 | 2
Pain in Pelvis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2
Dyspnea (Shortness of Breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated before the accrual goal was met as it was determined that the study lacked efficacy. Most patients did not reach 3 cycles of treatment in order to be evaluable for response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes